CLINICAL TRIAL: NCT04678596
Title: Comparison Of Different Orthodontic Aligner Systems Applied On Single Stage And Three Stage In Terms Of Comfort, Satisfaction, Treatment Effects And Duration
Brief Title: Comparison Of Different Orthodontic Aligner Systems Applied On Single Stage And Three Stage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ahmet Yağcı, Associate Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDH-2017-7774
Record Dates: First submitted 2019-09-30; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Tooth Crowding; Tooth; Lesion, White Spot Lesions
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EonAligner (Active Comparator): Patients in the EonAligner group were given a single thickness and hardness aligner and were asked to use the same it for 3 weeks.
  Interventions: Device: EonAligner
- Clearfix (Active Comparator): In the Clearfix group, the patients were given three different thickness and hardness aligner and they were asked to use each aligner for one week from soft to hard.
  Interventions: Device: Clearfix

INTERVENTIONS:
Device: EonAligner — EonAligner system is one stage system.
  Arms: EonAligner
Device: Clearfix — Clearfix system is three-stage system.
  Arms: Clearfix

SUMMARY:
Applying to the Orthodontics Department of the Faculty of Dentistry of Erciyes University for orthodontic treatment, a periodontally healthy 16-26 year-old periodontally healthy, non-congenital or congenital anomaly in the craniofacial region; 25 patients with class 1 orthodontic malocclusion with moderate permeability will be included in the study. The patients will be divided into 2 groups, and the first group of 12 patients will have single-stage aligner; The second group of 13 patients is planned to apply 3-stage aligner.

DETAILED DESCRIPTION:
It is planned to take lateral cephalometric radiography, panoramic radiography before and after the orthodontic treatment, and in addition to orthodontic model and photograph records before, during and after the treatment. Patient comfort and satisfaction will be evaluated by applying questionnaires to patients before treatment, immediately after starting treatment, 2 days later, 1 week later, 1 month later, 1 week before and after the treatment, and the effects of 2 different treatment methods on the patients will be evaluated according to the data obtained. QLF recordings are also taken at the beginning of treatment and at 3-month intervals, and the effects of single plaque use and 3 different plaque use on white spot lesion formation will be evaluated.

Hays Nance analysis will be used in the orthodontic models to determine the change in the amount of perplexity. In this way, tooth movement speeds can be determined. There are studies in the literature with single-stage transparent plates, but there are no studies with different-stage plates. In our study, which of the two different types of treatment is more comfortable on patients and affects the movement of teeth faster; In addition, the investigators plan to investigate which one has a low risk of white spot lesions on the teeth.

ELIGIBILITY:
Inclusion Criteria:

* No systemic disease
* Being healthy as periodontal.
* No smoking.
* No previous orthodontic treatment.
* Lack of congenital tooth deficiency
* Permanent dentition
* Class 1 malocclusion
* No clefts
* No extracted teeth

Exclusion Criteria:

* Orthodontic treatment history
* Missing tooth
* Poor oral hygiene
* Lack of cooperation

Ages: 16 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Actual)
Dates: Start 2017-12-06 (Actual); Primary Completion 2018-05-10 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Aesthetic and comfortable orthodontic treatment with aligner systems | 2 years
  Surveys
Comfortable orthodontic treatment with aligner systems | 2 years
  Visual Analog Score for pain

SECONDARY OUTCOMES:
Quality of life at orthodontic treatment with aligner systems | 2 years
  Physicians Global Assessment to measure quality of life
Evaluation of white spot lesion formation | 2 years
  rate of new white spot formation

OTHER OUTCOMES:
Evaluation of white spot lesion formation | 2 years
  rate of new white spot formation
Change of pain during treatment | 2 years
  measurement of pain level (grading system, VAS scoring)

CONTACTS AND LOCATIONS:
Overall Officials: meltem özsaygılı, Research Ass, Study Chair — Erciyes University Faculty of Dentistry
Locations (1):
- Erciyes University, Faculty of Dentistry, Department of Orthodontics University university, Kayseri, Melikgazi, Turkey (Türkiye)

REFERENCES:
- [Background] Yagci A, Korkmaz YN, Buyuk SK, Yagci F, Atilla AO. White spot lesion formation after treatment with full-coverage rapid maxillary expanders. Am J Orthod Dentofacial Orthop. 2016 Mar;149(3):331-8. doi: 10.1016/j.ajodo.2015.08.015. PMID 26926020
- [Background] Tufekci E, Dixon JS, Gunsolley JC, Lindauer SJ. Prevalence of white spot lesions during orthodontic treatment with fixed appliances. Angle Orthod. 2011 Mar;81(2):206-10. doi: 10.2319/051710-262.1. PMID 21208070
- [Result] Kim TW, Echarri P. Clear aligner: an efficient, esthetic, and comfortable option for an adult patient. World J Orthod. 2007 Spring;8(1):13-8. PMID 17373221
- [Result] Gorelick L, Geiger AM, Gwinnett AJ. Incidence of white spot formation after bonding and banding. Am J Orthod. 1982 Feb;81(2):93-8. doi: 10.1016/0002-9416(82)90032-x. PMID 6758594